CLINICAL TRIAL: NCT01596088
Title: A Multicenter, Open Label, Single-arm Study of KDX-0811(Dexrazoxane) in the Treatment of Accidental Extravasation of Anthracycline Anti-cancer Agents
Brief Title: A Phase I/II Study of KDX-0811(Dexrazoxane) in the Treatment of Accidental Extravasation of Anthracycline Anti-cancer Agents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: KDX1101
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Results first posted 2015-03-13 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Extravasations of Anthracycline Anti-cancer Agents
Keywords: Extravasation; Anthracyclines
MeSH Terms: interventions — Dexrazoxane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug: Dexrazoxane (Experimental): Dexrazoxane should be given once daily for 3 consecutive days. The dose is:
  Day 1: 1000 mg/m2, Day 2: 1000 mg/m2, Day 3: 500 mg/m2 (body surface area)
  Interventions: Drug: Dexrazoxane

INTERVENTIONS:
Drug: Dexrazoxane

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of KDX-0811(Dexrazoxane) in the treatment of accidental extravasation of anthracycline anti-cancer agents.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected to have been exposed to extravasation of anthracycline

Exclusion Criteria:

* Patients reasonably suspected to have been exposed to extravasation by other compounds than anthracyclines through the same IV access, e.g. vincristine, mitomycin, and vinorelbine, all of which may cause ulceration

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Primary Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuro Takei, Study Director — Kissei Pharmaceutical Co., Ltd.
Locations (1):
- Japan, Tokyo and Other Japanese City, Japan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexrazoxane
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dexrazoxane
Number analyzed (Participants) | 2
Age, Customized [Number; unit: participants]
  >=20 and <65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of participants experienced adverse events
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Dexrazoxane
Number analyzed (Participants) | 2
participants | 2

ADVERSE EVENTS:
Arm/Group | Dexrazoxane
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexrazoxane (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexrazoxane (N=2)
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Blood urea increased (Investigations) | 1
Blood creatinine increased (Investigations) | 2
Malaise (General disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Headache (Nervous system disorders) | 2
Hypersensitivity (Immune system disorders) | 1
Infusion site reaction (General disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
White blood cell count decreased (Investigations) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Blood cholesterol increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No